CLINICAL TRIAL: NCT03878030
Title: Effect of Nusinersen on Motor Function in Adult Patients With Spinal Muscular Atrophy Types 2 and 3
Brief Title: Effect of Nusinersen on Adults With Spinal Muscular Atrophy
Status: Completed | Type: Observational
Sponsor: Northwell Health (Other)
Responsible Party: Sponsor
Other Study IDs: 18-0149
Record Dates: First submitted 2019-03-10; First posted 2019-03-18 (Actual); Last update posted 2023-03-20 (Actual); Status verified 2023-03

CONDITIONS: Adult Spinal Muscular Atrophy
MeSH Terms: conditions — Muscular Atrophy, Spinal | interventions — nusinersen

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Subjects with spinal muscular atrophy types 2 and 3: Intrathecal nusinersen will be administered to all subjects per FDA approved label.
  Interventions: Drug: nusinersen

INTERVENTIONS:
Drug: nusinersen — Subjects will receive nusinersen and be observed with motor assessments for 24 months
  Other Names: Spinraza

SUMMARY:
Observational study of adult patients with spinal muscular atrophy types 2 and 3 receiving nusinersen

DETAILED DESCRIPTION:
Observational study to assess effects of nusinersen on motor function in adult patients with spinal muscular atrophy who are both ambulatory and non-ambulatory. Subjects will receive standard of care with nusinersen intrathecal injection and undergo baseline and every 6 month motor assessments and pulmonary function testing during the first two years of treatment with nusinersen.

ELIGIBILITY:
Inclusion Criteria:

* Genetically confirmed 5q SMA
* ability to access intrathecal space for nusinersen injection

Exclusion Criteria:

* Renal impairment
* thrombocytopenia
* inability to access intrathecal space by CT or flouro guided injection

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Study Population: The population to be studied are a homogenous group of adult subjects with 5q SMA seeking treatment with nusinersen. The subjects will have a broad phenotype spectrum of motor weakness including ability to ambulate, non-ambulatory and varying degrees of upper limb motor function and respiratory and swallow abilities, with some more affected and requiring invasive ventilation or NIV, and/or PEG tubes for nutrition.
Sampling Method: Probability Sample
Enrollment: 12 (Actual)
Dates: Start 2019-04-01 (Actual); Primary Completion 2021-07-13 (Actual); Study Completion 2021-07-13 (Actual)

PRIMARY OUTCOMES:
Change in quantitative motor function | Two years
  Primary Endpoint: Change from baseline to end of study in quantitative motor strength by dynamometry of upper limb muscles - shoulder abduction and elbow flexion/extension.
Change in upper limb motor function | Two years
  Change from baseline to end of study in upper limb module score
Change in 6 minute walk test in ambulatory patients | Two years
  Change in 6 minute walk test from baseline to end of study

SECONDARY OUTCOMES:
Change in pulmonary function by spirometry forced vital capacity (FVC) | Two years
  Change in FVC from baseline to end of study
Change in 10 meter walk test in ambulatory patients | Two years
  Change from baseline to end of study in the 10 meter walk test
Change in compound muscle action potential (CMAP) amplitude by nerve conduction velocity (NCV) criteria | Two years
  Change from baseline to end of study in CMAP amplitude of responses from median, ulnar and peroneal motor nerves
Change in pulmonary function by spirometry forced expiratory volume (FEV) | Two years
  Change from baseline to end of study in FEV

CONTACTS AND LOCATIONS:
Overall Officials: Anthony Geraci, MD, Principal Investigator — Northwell Health
Locations (1):
- Northwell Health Neuroscience, Great Neck, New York, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Finkel RS, Mercuri E, Darras BT, Connolly AM, Kuntz NL, Kirschner J, Chiriboga CA, Saito K, Servais L, Tizzano E, Topaloglu H, Tulinius M, Montes J, Glanzman AM, Bishop K, Zhong ZJ, Gheuens S, Bennett CF, Schneider E, Farwell W, De Vivo DC; ENDEAR Study Group. Nusinersen versus Sham Control in Infantile-Onset Spinal Muscular Atrophy. N Engl J Med. 2017 Nov 2;377(18):1723-1732. doi: 10.1056/NEJMoa1702752. PMID 29091570
- [Result] Mercuri E, Darras BT, Chiriboga CA, Day JW, Campbell C, Connolly AM, Iannaccone ST, Kirschner J, Kuntz NL, Saito K, Shieh PB, Tulinius M, Mazzone ES, Montes J, Bishop KM, Yang Q, Foster R, Gheuens S, Bennett CF, Farwell W, Schneider E, De Vivo DC, Finkel RS; CHERISH Study Group. Nusinersen versus Sham Control in Later-Onset Spinal Muscular Atrophy. N Engl J Med. 2018 Feb 15;378(7):625-635. doi: 10.1056/NEJMoa1710504. PMID 29443664